CLINICAL TRIAL: NCT00420693
Title: Interest of Using the Sevoflurane in the Prevention of Newborns Pain
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Dr Fabrice MICHEL, Assistance Publique Hopitaux De Marseille
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006/15
Record Dates: First submitted 2006-11-23; First posted 2007-01-11 (Estimated); Last update posted 2009-01-15 (Estimated); Status verified 2009-01

CONDITIONS: Pain Measurement; Newborn
MeSH Terms: interventions — Sevoflurane

INTERVENTIONS:
Drug: sevoflurane

SUMMARY:
The objective of this randomized and controlled study is to compare the sedation with sevoflurane inhalation versus non-nutritive sucking and sucrose administration to facilitate peripheral inserted central catheter insertion in a pediatric and neonatal intensive care. Main measurements concern success or failure of insertion, duration of procedure, movements of the baby, tolerance of treatments evaluated by, mean arterial pressure, heart rate, respiratory frequency and oxygen saturation.

ELIGIBILITY:
Inclusion Criteria:

* Infants born between the 28th and 41th weeks of gestation admitted in intensive care unit
* Patient requiring a mechanical ventilation or CPAP
* Patient requiring a KTEC
* Given consent

Exclusion Criteria:

* Contraindication to sévoflurane
* Patient already sedated with morphin and/or hypnotics
* Patient presenting neurologic troubles
* Patient enrolled in other study*
* Infant without legacy representant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-08; Primary Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Lasted realization of the gesture defined by delay between the first draining and the end of the bandage | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: fabrice michel, MD, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille CHU Nord, Marseille, BdR, France

REFERENCES:
- [Derived] Michel F, Vialet R, Hassid S, Nicaise C, Garbi A, Thomachot L, DI Marco JN, Lagier P, Martin C. Sevoflurane for central catheter placement in neonatal intensive care: a randomized trial. Paediatr Anaesth. 2010 Aug;20(8):712-9. doi: 10.1111/j.1460-9592.2010.03334.x. PMID 20546160